**PRINCIPAL INVESTIGATOR:** Christine Alewine, M.D., Ph.D.

STUDY TITLE: A Phase II Trial of the Superenhancer Inhibitor Minnelide

in Advanced Refractory Adenosquamous Carcinoma of

the Pancreas (ASCP)

STUDY SITE: NIH Clinical Center

Cohort: *Affected patient – Screening* 

Consent Version: 03/10/2023

#### WHO DO YOU CONTACT ABOUT THIS STUDY?

**Principal Investigator:** Christine Alewine, M.D., Ph.D.

#### KEY INFORMATION ABOUT THIS RESEARCH

This consent form describes a research study and is designed to help you decide if you would like to be a part of the research study.

You are being asked to take part in a research study at the National Institutes of Health (NIH). This section provides the information we believe is most helpful and important to you in making your decision about participating in this study. Additional information that may help you decide can be found in other sections of the document. Taking part in research at the NIH is your choice.

You are being asked to take part in this study because you have adenosquamous carcinoma of the pancreas (ASCP) or high suspicion for ASCP.

This consent is for "screening." Screening is the process to find out if you are eligible to take part in the treatment part of this study.

Participants in the treatment part of this study will receive a drug called Minnelide. The use of Minnelide in this study is considered investigational, which means that it has not been approved by the U.S. Food and Drug Administration (FDA) to treat ASCP. However, the FDA has given us permission to use Minnelide in this study.

There may be other drugs that may be used to treat your disease, and these can be prescribed/given by your regular cancer doctor, even if you are not in this study. The way in which treatment is given in this study and the side effects are not significantly different than if you were to receive standard care therapy.

If you decide to join this screening study, here are some of the most important things that you should know that will happen:

We will review your health history. We will confirm your cancer diagnosis.

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)

Version Date: 03/10/2023




- We will also do some basic tests to make sure you qualify for the trial. This will include physical exams, blood and urine tests, and tests to look at your heart function.
- Some of the tests have risks, including risks from blood samples and contrast with the imaging. We do not know which side effects you will experience.

There is no direct benefit to you from this part of the study. This screening part will help us decide if you are able to take part in the next step of this research study. You will have the benefit of seeing our NIH doctors to discuss your treatment. If you would like, we can share the results of these screening tests and notes with your personal physician.

The screening portion of this study will take between a few days and a week. If you move on to the treatment portion of the study, you may be in the study for several years depending on how you tolerate the treatment.

You are free to stop participating in the trial at any time. If you decide to stop, the study doctor may ask you to agree to certain tests to make sure it is safe for you to stop.

The remaining document will now describe the research study in more detail. This information should be considered before you make your choice. Members of the study team will talk with you about the information in this document. Some people have personal, religious, or ethical beliefs that may limit the kinds of medical or research interventions in which they would want to participate. Take the time you need to ask any questions and discuss this study with NIH staff, and with your family, friends, and personal health care providers.

#### IT IS YOUR CHOICE TO TAKE PART IN THE STUDY

You may choose not to take part in this study for any reason. If you join this study, you may change your mind and stop participating in the study at any time and for any reason. In either case, you will not lose any benefits to which you are otherwise entitled. However, to be seen at the NIH, you must be taking part in a study or are being considered for a study. If you do choose to leave the study, please inform your study team to ensure a safe withdrawal from the research.

#### WHY IS THIS STUDY BEING DONE?

The purpose of the treatment part of this research study is to see if Minnelide is an effective treatment for ASCP.

This part of the study is to determine if you are suited for the treatment part of this study.

You may not be eligible for our study for several reasons, such as the presence of certain other diseases, infections, or problems with your organ function.

#### WHAT WILL HAPPEN DURING THE STUDY?

Before you begin the study therapy, you will have several tests performed to check whether the study is suitable for you. This is called screening. Your doctor will review your medical history and the drugs that you are currently taking as well as the previous treatments you received for your disease to determine whether you can participate in this study.

Some of these tests or procedures are part of regular care and may be done even if you are not being considered to join the study. Most tests must be performed within 21 days before the start

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)




of treatment. If you have had some of these tests or procedures recently, they may or may not have to be repeated. Briefly, these tests include:

- Medical history: A complete review of your medical history, including obtaining information about your diagnosis and previous treatments, and reviewing information about your other conditions. If you have medical records from another clinic or hospital, you will be asked to get copies of these records, or your study doctor may be able to request them on your behalf. We will also collect information about your symptoms, any ongoing effects of prior treatment, and collect information about other medications you may be taking.
- Physical examination including weight and height, and vital signs.
- Performance status: an evaluation of your ability to perform everyday activities
- Electrocardiogram (ECG) to check your heart function.
- Computerized Tomography (CT) scan, magnetic resonance imaging (MRI), and/or brain scan.
- Lab blood and urine tests, to check for blood counts, organ function, and for signs of infection.
- Pregnancy test in women who can have children. Pregnant women will not be allowed on study.
- Test for hepatitis B and C
- Tissue from a tumor biopsy will be collected to confirm your cancer diagnosis. If tissue from a former biopsy is not available, you will be required to have a new biopsy to be reviewed.

#### HOW LONG WILL THE STUDY TAKE?

If you agree to take part in this study, the screening tests are expected to require about a week to be completed. After the evaluations are complete, we will determine if you are eligible to participate in the treatment portion of the study.

#### HOW MANY PEOPLE WILL PARTICIPATE IN THIS STUDY?

We plan to have approximately 55 people participate in this study at the NIH.

## WHAT ARE THE RISKS AND DISCOMFORTS OF BEING IN THE STUDY?

The primary risks or discomforts of participating in this screening are from complications caused by the tests and procedures. The following describes the most common risks of these tests and procedures. Your doctor or nurse will also discuss with you in detail any risks or discomforts of the procedures or test(s) you will be scheduled to undergo.

## **Risks from Study Procedures**

The following study procedures and treatments may have risks and cause discomfort while you participate on this study:

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)




#### **Blood draws**

Risks include temporary discomfort, pain, redness, bleeding, bruising, and swelling at the site where the needle is inserted, and/or very rarely inflammation/infection of the vein, which could require antibiotics. You may also experience dizziness, nausea, or rarely, fainting during blood taking. Please tell the study doctor if you do not feel well after having your blood drawn. We will collect up to 1 tablespoons of blood during the screening visit.

#### **Urine collection**

There is no risk related to urine collection.

## **Electrocardiogram (ECG)**

Some skin irritation can occur where the ECG/EKG electrodes are placed. Once the electrodes are placed, the test will begin, is completely painless, and generally takes less than a minute to perform. After the test, the electrodes are removed.

## **Imaging**

In addition to the radiation risks discussed below, CT scans may include the risks of an allergic reaction to the contrast. Participants might experience hives, itching, headache, difficulty breathing, increased heartrate and swelling.

#### Risks for MRI

Magnetic resonance imaging (MRI) uses a strong magnetic field and radio waves to take pictures of the body. We will obtain pictures of your chest, abdomen and pelvis for this study. The MRI scanner is a metal cylinder surrounded by a strong magnetic field. People are at risk for injury from the MRI magnet if they have some kinds of metal in their body. It may be unsafe for you to have an MRI scan if you have pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips (metal clips on the wall of a large artery), metal prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, tattoos, an implanted delivery pump, or shrapnel fragments. Welders and metal workers may have small metal fragments in the eye. You will be screened for these conditions before having any MRI scan. If you have a question about metal in your body, you should inform the staff. You will be asked to complete an MRI screening form before each MRI scan you have.

In addition, all magnetic objects (like watches, coins, jewelry, and credit cards) must be removed before entering the MRI scan room.

People with fear of confined spaces may become anxious during an MRI. Those with back problems may have back pain or discomfort from lying in the scanner. The noise from the scanner is loud enough to damage hearing, especially in people who already have hearing loss. Everyone having a research MRI scan will be fitted with hearing protection. If the hearing protection comes loose during the scan, you should let us know right away.

There are no known long-term risks of MRI scans.

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)




#### Risks from Gadolinium

During part of the MRI you will receive gadolinium, a contrast agent, through an intravenous (IV) catheter (small tube). It will be done for both research and medical purposes.

It is not known if MRI with contrast is completely safe for a developing fetus. Therefore, all women of childbearing potential will have a pregnancy test performed no more than 24 hours before each MRI scan with contrast. The scan will not be done if the pregnancy test is positive.

The risks of an IV catheter include bleeding, infection, or inflammation of the skin and vein with pain and swelling.

Mild symptoms from gadolinium infusion occur in fewer than 1% of those who receive it and usually go away quickly. Mild symptoms may include coldness in the arm during the injection, a metallic taste, headache, and nausea. In an extremely small number, fewer than one in 300,000 people, more severe symptoms have been reported including shortness of breath, wheezing, hives, and lowering of blood pressure. You should not receive gadolinium if you previously had an allergic reaction to it. You will be asked about such allergic reactions before gadolinium is given.

People with kidney disease are at risk for a serious reaction to gadolinium contrast called "nephrogenic systemic fibrosis (NSF)". This condition always involves the skin and can also involve the muscles, joints and internal organs. NSF has resulted in a very small number of deaths. A blood test of your kidney function may be done within the month before an MRI scan with gadolinium contrast. You will not receive gadolinium for a research MRI scan if your kidney function is below the safe level.

Most of the gadolinium contrast leaves the body in the urine. However, the FDA has issued a safety alert that indicates small amounts of gadolinium may remain in the body for months to years. The effects of the retained gadolinium are not clear. At this time, retained gadolinium has not been linked to health risks in people whose kidneys work well. Some types of gadolinium contrast drugs are less likely to remain in the body than others. In this study, we will use the gadolinium contrast drugs that are less likely to remain in the body.

# What are the risks related to pregnancy?

You may not participate in this study if you are pregnant. If you are able to become pregnant, we will perform a pregnancy test before exposing you to radiation. You must tell us if you may have become pregnant within the previous 14 days because the pregnancy test is unreliable during that time.

# What are the risks of radiation from being in the study?

During your participation in this part of the research study, you may be exposed to radiation from up to 1 CT scan. The amount of radiation exposure from these procedures is equal to approximately 1.3 rem. A rem is a unit of absorbed radiation.

Every day, people are exposed to low levels of radiation that come from the sun and the environment around them. The average person in the United States receives a radiation exposure of 0.3 rem per year from these sources. This type of radiation is called "background radiation." No one knows for sure whether exposure to these low amounts of radiation is harmful to your

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)




body.

The CT scan that you get in this study will expose you to the roughly the same amount of radiation as 4.3 years' worth of background radiation. Most of the time, this amount of extra radiation is not harmful to you. However, scientists believe that being exposed to too much radiation can cause harmful side effects. This could include getting a new cancer. We estimate that this could happen in about 1 out of every 1000 people who get a very large amount of extra radiation.

# WHAT ARE THE BENEFITS OF BEING IN THE STUDY?

You might not benefit from being in this study.

This part of the study is only for screening. However, you may gain clinical information about your disease or your organ function that will be helpful to your overall medical care. This testing may make you eligible to participate in this research study at the NIH. You will also have the benefit of a consultation with one of the NIH doctors to discuss your treatment, and, if you so desire, the results of these screening tests and procedures will be communicated to your personal physician.

## Are there any potential benefits to others that might result from the study?

In the future, other people might benefit from this study because of the knowledge gained from this therapeutic intervention for those eligible to receive it.

#### WHAT OTHER OPTIONS ARE THERE FOR YOU?

Before you decide whether or not to be in this study, we will discuss other options that are available to you. Instead of being in this study, you may choose not to be tested for eligibility or to have any other studies done.

#### DISCUSSION OF FINDINGS

## New information about the study

If we find out any new information that may affect your choice to participate in this study, we will get in touch with you to explain what we have learned. This may be information we have learned while doing this study here at the NIH or information we have learned from other scientists doing similar research in other places.

#### Return of research results

All of the clinical test results will be shared with you. We will discuss any findings that are abnormal with you. We can also share the findings of these screening evaluations with any medical provider that you wish to have this information.

#### EARLY WITHDRAWAL FROM THE STUDY

You will be removed from the study if:

• You are found not to be eligible for the study

You can stop taking part in the study at any time. However, if you decide to stop taking part in the study, we would like you to talk to the study doctor and your regular doctor first.

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)




# STORAGE, SHARING AND FUTURE RESEARCH USING YOUR SPECIMENS AND DATA

## Will your specimens or data be saved for use in other research studies?

As part of this study, we are obtaining specimens and data from you. We will remove all the identifiers, such as your name, date of birth, address, or medical record number and label your specimens and data with a code so that you cannot easily be identified. However, the code will be linked through a key to information that can identify you. We plan to store and use these specimens and data for studies other than the ones described in this consent form that are going on right now, as well as studies that may be conducted in the future. These studies may provide additional information that will be helpful in understanding ASCP, or other diseases or conditions. This could include studies to develop other research tests, treatments, drugs, or devices, that may lead to the development of a commercial product by the NIH and/or its research or commercial partners. There are no plans to provide financial compensation to you if this happens. Also, it is unlikely that we will learn anything from these studies that may directly benefit you.

I give permission for my coded specimens and data to be stored and used for future research as described above.

| Yes | No |
|----------|-----------------|
| Initials | <b>Initials</b> |

## Will your specimens or data be shared for use in other research studies?

We may share your coded specimens and data with other researchers. If we do, while we will maintain the code key, we will not share it, so the other researchers will not be able to identify you. They may be doing research in areas that are similar to this study or in other unrelated areas. These researchers may be at NIH, other research centers and institutions, or commercial entities.

I give permission for my coded specimens and data to be shared with other researchers and used by these researchers for future research as described above.

| Yes | No |
|----------|----------|
| Initials | Initials |

If you change your mind and do not want us to store and use your specimens and data for future research, you should contact the research team member identified at the top of this document. We will do our best to comply with your request but cannot guarantee that we will always be able to destroy your specimens and data. For example, if some research with your specimens and data has already been completed, the information from that research may still be used. Also, for

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17) File in Section 4:

File in Section 4: Protocol Consent (1) Version Date: 03/10/2023




example, if the specimens and data have been shared already with other researchers, it might not be possible to withdraw them.

In addition to the planned use and sharing described above, we might remove all identifiers and codes from your specimens and data and use or share them with other researchers for future research at the NIH or other places. When we or the other researchers access your anonymized data, there will be no way to link the specimens or data back to you. We will not contact you to ask your permission or otherwise inform you before we do this. We might do this even if you answered "no" to the above questions. If we do this, we would not be able to remove your specimens or data to prevent their use in future research studies, even if you asked, because we will not be able to tell which are your specimens or data.

NIH policies require that your clinical and other study data be placed in an internal NIH database that is accessible to other NIH researchers for future research. Usually, these researchers will not have access to any of your identifiers, such as your name, date of birth, address, or medical record number; and your data will be labeled with only a code. We cannot offer you a choice of whether your data to be placed in this database or not. If you do not wish to have your data placed in this database, you should not enroll in this study.

## How long will your specimens and data be stored by the NIH?

Your specimens and data may be stored by the NIH indefinitely.

## Risks of storage and sharing of specimens and data

When we store your specimens and data, we take precautions to protect your information from others that should not have access to it. When we share your specimens and data, we will do everything we can to protect your identity, for example, when appropriate, we remove information that can identify you. Even with the safeguards we put in place, we cannot guarantee that your identity will never become known or someone may gain unauthorized access to your information. New methods may be created in the future that could make it possible to re-identify your specimens and data.

#### **PAYMENT**

### Will you receive any type of payment for taking part in this study?

You will not receive any payment for taking part in this study.

#### REIMBURSEMENT

#### Will you receive reimbursement or direct payment by NIH as part of your participation?

On this study, the NCI will cover the cost for some of your expenses. Some of these costs may be paid directly by the NIH and some may be reimbursed after you have paid. The amount and form of these payments are determined by the NCI Travel and Lodging Reimbursement Policy. You will be given a summary of the policy which provides more information.

If your travel to the NIH Clinical Center (e.g. flight, hotel) is arranged and paid for by the NIH, the agency making the reservations and their representatives will have access to your identifiable information..

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)




#### **COSTS**

## Will taking part in this research study cost you anything?

NIH does not bill health insurance companies or participants for any research or related clinical care that you receive at the NIH Clinical Center.

- If some tests and procedures are performed outside the NIH Clinical Center, you may have to pay for these costs if they are not covered by your insurance company.
- Medicines that are not part of the study treatment will not be provided or paid for by the NIH Clinical Center.
- Once you have completed taking part in the study, medical care will no longer be provided by the NIH Clinical Center.

## **CONFLICT OF INTEREST (COI)**

The National Institutes of Health (NIH) reviews NIH staff researchers at least yearly for conflicts of interest. This process is detailed in a COI Guide. You may ask your research team for a copy of the COI Guide or for more information. Members of the research team who do not work for NIH are expected to follow these guidelines or the guidelines of their home institution, but they do not need to report their personal finances to the NIH.

Minneamrita Therapeutics is providing Minnelide for this study to NIH without charge. No NIH employee involved in this study receives any payment or other benefits from Minneamrita Therapeutics.

#### CLINICAL TRIAL REGISTRATION AND RESULTS REPORTING

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

## CONFIDENTIALITY PROTECTIONS PROVIDED IN THIS STUDY

Some of your health information, and/or information about your specimen, from this study will be kept in a central database for research. Your name or contact information will not be put in the database. Your test results will be identified by a unique code and the list that links the code to your name will be kept separate from your sample and health information. Your information may be given out if required by law. For example, certain states require doctors to report to health boards if they find a disease like tuberculosis. However, the researchers will do their best to make sure that any information that is released will not identify you.

## Will your medical information be kept private?

We will do our best to make sure that the personal information in your medical record will be kept private. However, we cannot guarantee total privacy. Organizations that may look at and/or copy your medical records for research, quality assurance, and data analysis include:

- The NIH and other government agencies, like the Food and Drug Administration (FDA), which are involved in keeping research safe for people.
- National Institutes of Health Intramural Institutional Review Board
- The study Sponsor, Center for Cancer Research, or their agent(s)

#### PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)




 Qualified representatives from Minneamrita Therapeutics, the pharmaceutical company who produces Minnelide.

The researchers conducting this study and the NIH follow applicable laws and policies to keep your identifying information private to the extent possible. However, there is always a chance that, despite our best efforts, your identity and/or information about your participation in this research may be inadvertently released or improperly accessed by unauthorized persons.

In most cases, the NIH will not release any identifiable information collected about you without your written permission. However, your information may be shared as described in the section of this document on sharing of specimens and data, and as further outlined in the following sections.

Further, the information collected for this study is protected by NIH under a Certificate of Confidentiality and the Privacy Act.

## **Certificate of Confidentiality**

To help us protect your privacy, the NIH Intramural Program has received a Certificate of Confidentiality (Certificate). With this certificate, researchers may not release or use data or information about you except in certain circumstances.

NIH researchers must not share information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings, for example, if requested by a court.

The Certificate does not protect your information when it:

- 1. is disclosed to people connected with the research, for example, information may be used for auditing or program evaluation internally by the NIH; or
- 2. is required to be disclosed by Federal, State, or local laws, for example, when information must be disclosed to meet the legal requirements of the federal Food and Drug Administration (FDA);
- 3. is for other research;
- 4. is disclosed with your consent.

The Certificate does not prevent you from voluntarily releasing information about yourself or your involvement in this research.

The Certificate will not be used to prevent disclosure to state or local authorities of harm to self or others including, for example, child abuse and neglect, and by signing below you consent to those disclosures. Other permissions for release may be made by signing NIH forms, such as the Notice and Acknowledgement of Information Practices consent.

## **Privacy Act**

The Federal Privacy Act generally protects the confidentiality of your NIH medical information that we collect under the authority of the Public Health Service Act. In some cases, the Privacy Act protections differ from the Certificate of Confidentiality. For example, sometimes the Privacy Act allows release of information from your record without your permission, for example, if it is requested by Congress. Information may also be released for certain research purposes with due consideration and protection, to those engaged by the agency for research purposes, to certain federal and state agencies, for HIV partner notification, for infectious disease or abuse or neglect

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1) Version Date: 03/10/2023

Dags 10 of 12




reporting, to tumor registries, for quality assessment and medical audits, or when the NIH is involved in a lawsuit. However, NIH will only release information from your medical record if it is permitted by both the Certificate of Confidentiality and the Privacy Act.

#### POLICY REGARDING RESEARCH-RELATED INJURIES

The NIH Clinical Center will provide short-term medical care for any injury resulting from your participation in research here. In general, no long-term medical care or financial compensation for research-related injuries will be provided by the NIH, the NIH Clinical Center, or the Federal Government. However, you have the right to pursue legal remedy if you believe that your injury justifies such action.

# PROBLEMS OR QUESTIONS

| If you have any problems or question | s about this study, or about your rights as a researc | h |
|---|---|---|
| participant, or about any research-relat | ted injury, contact the Principal Investigator, Christin | le |
| Alewine, | You may also call the NIH Clinical Center | er |
| Patient Representative at 3 | or the NIH Office of IRB Operations at | if |
| you have a research-related complaint or | concern. | |

#### CONSENT DOCUMENT

Please keep a copy of this document in case you want to read it again.

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17) File in Section 4: Protocol Consent (1) Version Date: 03/10/2023




| Signature of Research Participant | Print Name of Researce<br>Participant | ch Date |
|---|---|---|
| Investigator: | | |
| Signature of Investigator | Print Name of Investigator | Date |
| Witness should sign below if either: | cess has been used to enroll a n | on-English sneaking |
| subject or | full consent has been used to enro | |
| subject or 2. An oral presentation of the subject | | |
| subject or 2. An oral presentation of the subject Signature of Witness NIH ADMINISTRATIVE SECTIO | Print Name of Witness | Il a blind or illiterate Date |
| subject or 2. An oral presentation of the subject Signature of Witness NIH ADMINISTRATIVE SECTION INTERPRETER: | Print Name of Witness | Date DING THE USE OF |
| subject or 2. An oral presentation of the subject Signature of Witness NIH ADMINISTRATIVE SECTIO AN INTERPRETER: An interpreter, or other individual | Print Name of Witness N TO BE COMPLETED REGAR ual, who speaks English and the pent and served as a witness. The interest of the complete served as a witness. | Date Date Date Darticipant's preferred |
| subject or 2. An oral presentation of the subject Signature of Witness NIH ADMINISTRATIVE SECTION INTERPRETER: An interpreter, or other individual language facilitated the administration of informed consent may not also serve as the witness. | Print Name of Witness N TO BE COMPLETED REGAR ual, who speaks English and the pent and served as a witness. The interest of the complete served as a witness. | Date |
| Signature of Witness NIH ADMINISTRATIVE SECTION AN INTERPRETER: An interpreter, or other individual language facilitated the administration of informed conseconsent may not also serve as the witness. | Print Name of Witness N TO BE COMPLETED REGAR ual, who speaks English and the pent and served as a witness. The inness. ual, who speaks English and the pent and served as a witness. | Date Darticipant's preferred investigator obtaining Darticipant's preferred |

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


